CLINICAL TRIAL: NCT04015141
Title: An Open-Label Study With Extension Phase to Evaluate the Efficacy and Safety of Perampanel Administered as an Adjunctive Therapy in Pediatric Subjects (Age 1 Month to Less Than 18 Years) With Childhood Epilepsy
Brief Title: A Study to Evaluate Efficacy and Safety of Perampanel Administered as an Adjunctive Therapy in Pediatric Participants With Childhood Epilepsy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-G000-236; 2018-004456-38 (EudraCT Number)
Record Dates: First submitted 2019-05-27; First posted 2019-07-10 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Epileptic Syndrome; Partial-onset Seizures
Keywords: Partial-onset seizures; Pediatric epileptic syndrome; Epilepsy; Childhood epilepsy; Epilepsy in children; Refractory seizures; Inadequately controlled seizures; E2007; Fycompa; Perampanel
MeSH Terms: conditions — Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Perampanel (Experimental): Participants aged 1 month to less than 18 years with pediatric epileptic syndrome (Cohort 1) or aged 1 month to less than 2 years with POS (Cohort 2) will receive perampanel oral suspension or perampanel tablets, once daily up to 56 weeks.
  Interventions: Drug: Perampanel Oral Suspension; Drug: Perampanel Tablet

INTERVENTIONS:
Drug: Perampanel Oral Suspension — Perampanel oral suspension.
  Other Names: E2007; Fycompa
Drug: Perampanel Tablet — Perampanel tablet.
  Other Names: E2007; Fycompa

SUMMARY:
The purpose of the study is to evaluate the efficacy of perampanel as measured by the 50 percent (%) responder rate during the maintenance period of the core study for seizure frequency in participants with pediatric epileptic syndrome (Cohort 1) and partial-onset seizures (POS) (Cohort 2).

DETAILED DESCRIPTION:
This study will consist of a Core Study, Extension Phase A and Extension Phase B.

1. Core Study will consist of the following 2 phases: Pretreatment (4 weeks screening or baseline period) and Treatment Period. The Treatment Period (23 weeks) of Core study include Titration period (10 weeks) and Maintenance period (13 weeks).
2. Extension Phase A will consist of a Treatment Period (33 weeks) and a Follow-up Period (4 weeks). All participants who will complete the Core Study will be eligible to participate in Extension Phase A of the study.
3. Extension Phase B will only be for participants who reside in countries where perampanel (oral tablets or oral suspension) is not commercially available or an extended access program (EAP) is not yet implemented, participants have completed Extension Phase A, and who, in the opinion of the investigator, will continue to benefit from treatment with perampanel.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants. Cohort 1: age 1 month to less than 18 years; Cohort 2: age 1 month to less than 2 years at the time of informed consent/assent. Participants below the age of 1 year must have been at least 36 weeks of gestational age at birth.
* Have a diagnosis of epilepsy with a pediatric epileptic syndrome (Cohort 1) or epilepsy with POS with or without secondary generalization (Cohort 2).
* Have had equal or greater than 4 seizures over the 4-week interval prior to enrollment visit.
* Absence of any progressive cause of epilepsy that has been confirmed clinically or based on brain imaging (example, magnetic resonance imaging [MRI] scan or computed tomography [CT] or ultrasound [for less than 1 year old]).
* Currently maintained on stable doses of 1 to a maximum of 4 approved antiepileptic drugs (AEDs). A prescription medical marijuana (including products containing cannabidiol) is counted as 1 of the maximum of 4 allowed AEDs; however, it cannot be the only concomitant AED if this product is not an approved AED in the country where the study site is located. Doses must be stable for at least 4 weeks (at least 2 weeks for participant less than [<] 6 months old) before Visit 1/Baseline or screening; only 1 enzyme-inducing antiepileptic drug (EIAED) (defined as carbamazepine, phenytoin, oxcarbazepine, or eslicarbazepine) out of the maximum of 4 AEDs is allowed.

Exclusion Criteria:

* Current or history of pseudo-seizures (psychogenic nonepileptic seizures) within approximately 5 years before screening visit.
* Have a history of status epilepticus that required hospitalization within 6 months before screening visit.
* Have an unstable psychiatric diagnosis that may confound participant's ability to participate in the study or that may prevent completion of the protocol specified tests (example, significant suicide risk, including suicidal behavior and ideation within 6 months before screening visit 1, current psychotic disorder, acute mania).
* Any suicidal ideation with intent with or without a plan within 6 months before enrollment visit (answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the C-SSRS) in participants aged 6 and above or based on the opinion of the Investigator for participants less than 6 years.
* Are scheduled or confirmed or both to have epilepsy surgery within 6 months after screening visit; however, those who have previously documented "failed" epilepsy surgery will be allowed.
* Have a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors.
* Benzodiazepines for any indications other than epilepsy (example, anxiety/sleep disorders) prohibited from 1 month before Visit 1/Baseline or screening and during the study. Benzodiazepines for seizure control and as rescue medication are allowed.
* A vagal nerve stimulator (VNS), responsive neurostimulator (RNS), or deep brain stimulator (DBS) implanted less than 5 months before screening visit or changes in parameter less than 4 weeks before screening visit (or thereafter during the study).
* Use of perampanel within 30 days before screening visit, or perampanel was discontinued due to adverse reactions (perampanel-related) or lack of efficacy in case of previous exposure.
* Weight less than 4.0 kilogram (kg) at Visit 1 (Baseline or screening).

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2027-04-06 (Estimated); Study Completion 2027-12-23 (Estimated)

PRIMARY OUTCOMES:
Proportion of 50% Responders For All Seizures During the Maintenance Period of Core Study | Week 10 to Week 23
  A response of 50% will be defined as a decrease in 28-day seizure frequency of equal or greater than 50% compared to baseline seizure frequency.

SECONDARY OUTCOMES:
Proportion of 50% Responders During Treatment Period of Core Study and Extension Phase A | Treatment Period of Core Study and Extension Phase A: Week 0 to Week 56
  A response of 50% is defined as a decrease in 28-day seizure frequency of equal or greater than 50% compared to baseline seizure frequency.
Proportion of 25% and 75% Responders for all Seizures, During Maintenance Period of Core Study and During Treatment Period of Core Study and Extension Phase A | Maintenance Period of Core study: Week 10 to Week 23; Treatment Period of Core Study and Extension Phase A: Week 0 to Week 56
  A response of 25% is defined as a decrease in 28-day seizure frequency of equal or greater than 25% compared to baseline seizure frequency. 75% response is defined as a decrease in 28-day seizure frequency of equal or greater than 75% compared to baseline seizure frequency.
Proportion of Participants Who Are Seizure-Free During the Maintenance Period of Core Study and During the Treatment Period of Core Study and Extension Phase A | Maintenance Period of Core study: Week 10 to Week 23; Treatment Period of Core Study and Extension Phase A: Week 0 to Week 56
Change From Baseline in Seizure Frequency For All Seizures During the Treatment Period of Core Study and During the Treatment Period of Core Study and Extension Phase A | Baseline, Treatment Period of Core study: Week 23, Treatment Period of Core Study and Extension Phase A: Week 56
Percent Change From Baseline in Seizure Frequency For All Seizures During the Treatment Period of Core Study and During the Treatment Period of Core Study and Extension Phase A | Baseline, Treatment Period of Core study: Week 23, Treatment Period of Core Study and Extension Phase A: Week 56
Clinical Global Impression of Change (CGIC) at the End of the Treatment Period of Core Study and at the End of Extension Phase A | Treatment Period of Core Study: Week 23, Extension Phase A: Week 56
  Assessment of disease severity will utilize the CGIC scale at end of treatment to evaluate participant's change in disease status since initiation of treatment. The CGIC is a 7-point scale that measures a physician's global impression of a participant's clinical condition. Scale ranges from 1 to 7 with lower scores indicating improvement (1=very much improved, 2=much improved, 3=minimally improved), higher scores indicating worsening (5=minimally worse, 6= much worse, 7=very much worse), and a score of 4 indicating no change.
Subject Global Impression of Change (SGIC) at the End of the Treatment Period of Core Study and at the End of Extension Phase A | Treatment Period of Core Study: Week 23, Extension Phase A: Week 56
  SGIC is a 7-Point scale that provides a participant-determined summary measure of change from baseline of participant's status. Scale ranges from 1 to 7 with lower scores indicating improvement (1=very much improved, 2=much improved, 3=minimally improved), higher scores indicating worsening (5=minimally worse, 6= much worse, 7=very much worse), and a score of 4 indicating no change.
Change From Baseline in the Cognitive Drug Research (CDR) Parameter at the End of the Treatment Period of Core Study and at the End of Extension Phase A | Baseline, Treatment Period of Core Study: Week 23, Extension Phase A: Week 56
  The CDR System Global Cognition Score (cognitive test battery) is derived from 5 CDR System domain scores, also called factor scores: Power of Attention, Continuity of Attention, Quality of Episodic Memory, Quality of Working Memory, and Speed of Memory. The CDR assessment and Child Behavior Checklist (CBCL) will be administered to participants 6 years and over and 2 years and over, respectively, using an age-appropriate version to assess cognitive function and behavior.
Change from Baseline in CBCL Parameters at the End of the Treatment Period of Core Study and at the End of Extension Phase A | Baseline, Treatment Period of Core Study: Week 23, Extension Phase A: Week 56
  The CBCL is a questionnaire to assess behavioral and emotional problems in children as reported by the primary caregiver. It is standardized to evaluate maladaptive behavioral and emotional problems in ages 1.5 to 5 years (CBCL 1.5/5) or 6 to 18 years (CBCL). The CBCL examines three domains (Social Functioning, Mood and Anxiety Symptoms, and Externalizing Symptoms) by assessing 140 problem items that describe specific behavioral and emotional problems. Respondents indicate how accurately the statements describe the child by selecting from options on a 3-point Likert-type scale (0=Not True, 1= Somewhat or Sometimes True, or 2=Very True or Often True).
Change from Baseline in Lafayette Grooved Pegboard Test (LGPT) Parameters at the End of the Treatment Period of Core Study and at the End of Extension Phase A | Baseline, Treatment Period of Core Study: Week 23, Extension Phase A: Week 56
  LGPT measures visuomotor skills. This test is a manipulative dexterity test that consist of a metal matrix of 25 holes with randomly positioned slots. Participants require to insert 10 grooved pegs into the holes. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. The task is timed and the scores are the time taken for the participant to complete all 10 pegs for each hand. If the test cannot be completed within 300 seconds, 300 seconds are recorded for the time. An increase in score (longer time) indicates worsening of visuomotor skills.
Change from Baseline in Growth and Development Parameter - Height | Baseline, Treatment Period of Core Study: Week 23; Extension Phase A: Weeks 28, 40, and 56
Change from Baseline in Growth and Development Parameter - Weight | Baseline, Treatment Period of Core Study: Weeks 2, 5, 8, 10, 14, 18 and 23; Extension Phase A: Weeks 28, 40, 56, and 60
Change from Baseline in Growth and Development Parameter - Free Triiodothyronine (fT3) and Free Thyroxine (fT4) Levels in Blood | Baseline, Treatment Period of Core Study: Week 23, Extension Phase A: Week 56
Change from Baseline in Growth and Development Parameter - Thyroid-Stimulating Hormone (TSH) Levels in Blood | Baseline, Treatment Period of Core Study: Week 23, Extension Phase A: Week 56
Change from Baseline in Growth and Development Parameter - Insulin Like Growth Factors (IGF)-1 | Baseline, Treatment Period of Core Study: Week 23, Extension Phase A: Week 56
Change from Baseline in Growth and Development Parameter- Sexual Maturation Assessed by Tanner Staging | Baseline, Treatment Period of Core Study: Week 23, Extension Phase A: Week 56
  Sexual maturation including pubic hair growth (both sexes), genital (males only) and breast (females only) development of participants will be assessed using Tanner Staging.
Proportion of Participants with any Treatment-Emergent Reports of Suicidal Ideation and Behavior on the Columbia-Suicide Severity Rating Scale (C-SSRS) and Intensity of These Behaviors Assessed using C-SSRS Scores | Treatment period of Core Study: Weeks 0, 2, 5, 8, 10, 14, 18, and 23; Extension Phase A: Weeks 28, 46, 56 and 60
  C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS is used to assess whether participant experienced SI (1:wish to be dead; 2:non-specific active suicidal thoughts; 3:active SI with any methods (not plan) without intent to act; 4:active SI with some intent to act, without specific plan; 5:active SI with specific plan and intent) and suicidal behavior (6:actual attempt; 7:interrupted attempt; 8:aborted attempt; 9:preparatory acts or behavior; 10:suicidal behavior). An assessment of SI and behavior using the C-SSRS will be performed throughout the study for participants aged 6 years and above at the time of consent. In participants younger than 6 years, SI and behavior will be monitored based upon clinical impression.
Change from Baseline in Number of Seizures Recorded on Electroencephalogram (EEG) at the End of the Treatment Period of Core Study and at the End of Extension Phase A | Baseline, End of the Treatment Period of Core Study: Week 23, End of Extension Phase A: Week 56
Number of Participants with at Least One Treatment Emergent Adverse Event (TEAE) and Serious Adverse Event (SAE) | From date of first dose of perampanel up to 28 days after the last dose of perampanel (Week 60)
Number of Participants with Treatment Emergent Markedly Abnormal Laboratory Values | From date of first dose of perampanel up to Week 60
Number of Participants with Clinically Notable Vital Sign Results | From date of first dose of perampanel up to 28 days after the last dose of perampanel (Week 60)
  Vital sign measurements include systolic and diastolic blood pressure [millimeters of Mercury (mmHg)], pulse (beats per minute), respiratory rate (per minute), temperature (degree centigrade), and weight (kilogram).
Number of Participants with Clinically Significant Abnormal Electrocardiograms | From date of first dose of perampanel up to Week 60

CONTACTS AND LOCATIONS:
Locations (49):
- United States (22):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Center For Neurosciences, Tucson, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Nemours Foundation Alfred Dupont Children's Hospital, Wilmington, Delaware
  - Nicklaus Children's Hospital, Miami, Florida
  - Pediatric Neurology PA, Orlando, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - PANDA Neurology, Atlanta, Georgia
  - Meridian Clinical Research-(Savannah Georgia), Savannah, Georgia
  - Children's Hospital of Michigan, Detroit, Michigan
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Wake Forest Baptist Medical Center - PPDS, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Child Neurology Consultants of Austin, Austin, Texas
  - Road Runner Research Ltd, San Antonio, Texas
  - Children's Specialty Group, Norfolk, Virginia
  - Children's Hospital of Richmond at VCU - CHoR-PIN, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Belgium (6):
  - Centre Neurologique William Lennox, Ottignies, Brabant Wallon
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - H�pital Universitaire des Enfants Reine Fabiola, Brussels, Brussels Capital
  - UZ Brussel, Brussels, Brussels Capital
  - UZ Gent, Ghent, Oost-Vlaanderen
  - H�pital Erasme, Anderlecht
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Plzen, Pilsen
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus N, Central Jutland
  - Regionshospitalet Randers, Randers
- France (6):
  - Hopitaux de La Timone, Marseille, Bouches-du-Rhone
  - H�pital Pellegrin-Enfants, Bordeaux
  - Hopital Necker, Paris
  - Hopitaux de Paris CHU Hopital Robert Debre - Inserm U676, Paris
  - CHRU Rennes, Rennes
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Germany (4):
  - Universit�tsklinikum Freiburg, Freiburg im Breisgau
  - Universit�tsklinikum Jena, Jena
  - Dr. Von Haunersches Kinderspital, Munich
  - Kleinwachau S�chsisches Epilepsiezentrum Radeberg Gemeinn�tzige Gmbh, Radeberg
- Spain (6):
  - Centro Medico Teknon � Grupo Quironsalud, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital General Universitario Gregorio Mara�on, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - CHUS � H. Clinico U. de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio - PPDS, Seville

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.